CLINICAL TRIAL: NCT01329211
Title: Needs Assessment Evaluating Quality of Life Issues for Gastroparesis Patients and Caregivers
Status: Terminated | Type: Observational
Why Stopped: PI left institution,replacement PI not able to do study.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 693-2009
Record Dates: First submitted 2011-03-24; First posted 2011-04-05 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Quality of Life
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastroparesis Patients
- Gastroparesis Patients' Caregivers

SUMMARY:
The project will involve conducting a Needs Assessment for Gastroparesis patients and their caregivers with the goal of identifying quality of life issues associated with this disease. Identifying these issues will ameliorate management and support systems for gastroparesis currently existent in the community and, hopefully, provide information for the establishment of more resources to assist the patients and their families.

DETAILED DESCRIPTION:
This project will involve: a) distributing questionnaires to up to 200 participants (100 patients and 100 caregivers) at the Shands Gastrointestinal clinic and b) focus groups including patients, medical provider, and the clinic case manager. The questionnaires will provide information on the relative effect of gastroparesis on the quality of life of the patients and their caregivers. Assessment of this needs assessment will then help identify areas of potential resource improvement and mobilization to provide support for the patients and their family members.

ELIGIBILITY:
Inclusion Criteria:

* Gastroparesis patients at the GI clinic of Shands Hospital at the University of Florida
* Caregivers to Gastroparesis patients at the GI clinic of Shands Hospital at the University of Florida

Exclusion Criteria:

* Inability to fill out the questionnaires by any cause

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The research plan involves reviewing patient records to identify potential subjects. Questionnaires will be distributed to gastroparesis patients and their caregivers during their visit to the GI clinic at the day of enrollment and at six-month intervals for a two-year follow-up period, after informed consent has been obtained. Patients and caregivers will also be recruited by telephone. Gastroparesis patients, who have an established patient-physician relationship with Dr. Sultan, will be contacted by telephone in order to inquire about their interest in participating in the study. The details of the study, including the questionnaires, risks, and potential benefits will be discussed over the phone. Then, if patients and/or their caregivers are willing to participate in the study, the informed consent forms and the questionnaires will be mailed to them with a posted envelope to be returned to Dr. Sultan by mail.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Score in a Quality of life assessment Questionnaire | During the clinicial visit at the day of enrollment(Day 1)

SECONDARY OUTCOMES:
Score in a Quality of life assessment Questionnaire | 1st follow-up, at 6 months from Date of enrollment
Score in a Quality of life assessment Questionnaire | 2nd follow-up, at 12 months from date of enrollment
Score in a Quality of life assessment Questionnaire | 3rd follow-up, at 18 months form date of enrollment
Score in a Quality of life assessment Questionnaire | 4th(last) follow-up, At 24 months form date of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Sultan, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States